CLINICAL TRIAL: NCT05729100
Title: The Effects of Preoperative Oral Carbohydrate-electrolyte Solution Compared to Standard Clear Fluid on Metabolic Responses, Preoperative Anxiety and Postoperative Complications in Paediatric Patients
Brief Title: The Effects of Carbohydrate-electrolyte Solution on Metabolic Responses in Paediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Principle Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes210
Record Dates: First submitted 2023-01-15; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Fasting
Keywords: preoperative fasting; carbohydrate; metabolic response; paediatrics; preoperative anxiety; post operative nausea and vomiting; emergence delirium; insulin resistance; HOMA-IR; Interleukin-6
MeSH Terms: conditions — Fasting; Vomiting; Emergence Delirium; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral carbohydrate-electrolyte solution (Experimental): The intervention group who will receive 50 ml/kg of oral solution containing carbohydrate-electrolyte
  Interventions: Other: Oral carbohydrate-electrolyte solution
- Standard clear fluid (Sham Comparator): The control group who will receive 50 ml/kg of clear fluid (i.e. water; which does not contain carbohydrate-electrolyte)
  Interventions: Other: Control

INTERVENTIONS:
Other: Oral carbohydrate-electrolyte solution — Oral solution containing 10% glucose and electrolyte (in every 300 ml of fluid (contains 30 gr dextrose, 150 mg Natrium chloride, 366 mg Kalium chloride)
  Arms: Oral carbohydrate-electrolyte solution
Other: Control — Standard clear fluid (water)
  Arms: Standard clear fluid

SUMMARY:
The aim of this study is to evaluate the effects of oral administration of carbohydrate-electrolyte-containing fluid, compared to standard clear fluid during preoperative fasting on metabolic responses, preoperative anxiety and postoperative complications in paediatric patients. Subjects will be randomly allocated into 2 groups: the intervention group will receive carbohydrate- electrolyte fluid whilst the control group will receive clear fluid. Both groups will receive 50 ml/kg of their designated fluid one day prior to surgery, and are allowed to consume the fluid gradually until 1 hour before the induction of anaesthesia. Prior to induction, preoperative anxiety will be assessed. Metabolic responses will be assessed through the degree of insulin resistance (using the Homeostatic Model Assessment for Insulin Resistance - HOMA-IR) and inflammatory cytokine (Interleukin-6) level. The metabolic responses will be evaluated after the induction of anaesthesia and 24 hours following the surgery. Preoperative anxiety will be assessed before the surgery using the Modified Yale Preoperative Anxiety Scale Short Form (mYPAS-SF). Immediate post operative complications such as post operative nausea and vomiting (PONV), emergence delirium and postoperative pain will be assessed in the recovery room.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of oral administration of carbohydrate-electrolyte-containing fluid, compared to standard clear fluid during preoperative fasting on metabolic responses, preoperative anxiety and postoperative complications in paediatric patients. Metabolic responses will be assessed through the degree of insulin resistance (using the Homeostatic Model Assessment for Insulin Resistance - HOMA-IR) and inflammatory cytokine (Interleukin-6) level. The metabolic responses will be evaluated after the induction of anaesthesia and 24 hours following the surgery. Preoperative anxiety will be assessed before the surgery using the Modified Yale Preoperative Anxiety Scale Short Form (mYPAS-SF). Immediate post operative complications such as post operative nausea and vomiting (PONV), emergence delirium and postoperative pain will be assessed in the recovery room. This study is a single-blinded randomised controlled trial. Subjects will be randomly allocated into 2 groups: the intervention group will receive carbohydrate-electrolyte fluid whereas the control group will receive clear fluid. Both groups will receive 50 ml/kg of their designated fluid one day prior to surgery, and are allowed to consume the fluid gradually since the fluid is given (approximately 12 hours before the surgery) until 1 hour before induction of anaesthesia. The fluid used in this study will be prepared by the Pharmacy Department, independent from the research team, in which the randomization and which fluid given to patients remain concealed from the primary research team.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 month - 12 years old
* Patients with physical status according to American Society of Anesthesiologists (ASA) 1 or 2
* Patients undergoing surgery with general anesthesia with or without regional anesthesia
* Has a relatively good enteral tolerability

Exclusion Criteria:

* Patients with endocrine abnormalities
* Patients requiring Pediatric intensive care unit (PICU) for post operative care and is likely to remain intubated following the end of the surgery
* Patients who receive antiemetic therapy within 24 hours before the surgery
* Patients undergoing cardiac surgery or neurosurgery

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 24 hours
  Insulin resistance will be evaluated using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), which is a model to estimate insulin sensitivity based on the ratio of insulin and blood glucose. The calculation of the HOMA-IR model uses the formula : HOMA-IR = insulin level (microIU/ml) x blood glucose level (mmol/L) / 22.5
  Insulin resistance will be evaluated after the induction of anesthesia, and 24 hours following the operation. Since HOMA-IR is a ratio that requires insulin and blood glucose level, the insulin level (microIU/ml) and the blood glucose level (mmol/L) will also be evaluated after the induction, and 24 hours following the operation. A higher HOMA-IR ratio represents an increased level of insulin resistance.
Interleukin-6 | 24 hours
  The level of interleukin-6 (pg/dl) in this study is evaluated to reflect the degree of body response to surgical trauma. It will be measured after the induction of anesthesia, and 24 hours after surgery. A higher interleukin-6 level indicates a higher inflammatory reaction following surgical trauma.

SECONDARY OUTCOMES:
Preoperative anxiety | 1 hour
  Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety - Short Form Scale. The scale incorporates 4 parameters to be assessed, the lowest score is 22.9 and the highest score is 61.45. The score below 61.45 is considered 'low anxiety' level, while the score at or more than 61.45 is considered 'high anxiety' level. This scale will be assessed when the patient arrived in the preparation room, before going to the operating room.
Post operative nausea and vomiting | 1 hour
  The incidence of post operative nausea and vomiting will be documented in a yes or no fashion. The post operative nausea and vomiting will be assessed after surgery in the recovery room.
Emergence Delirium | 1 hour
  The incidence of emergence delirium will be evaluated using the Paediatric Anaesthesia Emergence Delirium score. Emergence delirium will be assessed right after the surgery when the patient is in the recovery room. The lowest score is 0, the highest is 20. A higher score indicates a higher possibility for the occurrence of emergence delirium. The score of more than 12 is considered positive for the occurrence of emergence delirium.
Postoperative pain | 1 hour
  The postoperative pain will be assessed after the surgery in the recovery room using the Visual Analogue Scale. The score ranges from 0 (no pain) to 10 (worst pain). A higher score indicates a more severe pain.
  For the preverbal children who might be difficult to communicate the pain, the Face, Legs, Activity, Cry, Consolability (FLACC) scale will be used. This study uses the FLACC score for children younger than 7 years old. The FLACC score ranges from 0-10, the higher the score represent the more severe the pain might be.

CONTACTS AND LOCATIONS:
Locations (1):
- Ciptomangun Kusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No